CLINICAL TRIAL: NCT04594837
Title: Portable Ankle Robotics to Reverse Foot Drop After Stroke
Brief Title: Ankle Robotics After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NextStep Robotics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1 U44 111076-01
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Foot Drop; Stroke; Hemiparesis
MeSH Terms: conditions — Peroneal Neuropathies; Stroke; Paresis | interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PTR (Physical Therapy while wearing Robot group) (Phase II) (Experimental): Subjects receive 18 one-hour PT training sessions over 9 weeks while wearing the robot initially parameterized to individual deficit severity. Subjects perform over-ground mobility tasks of increasing challenge with robotic assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Interventions: Device: PTR Physical Therapy while wearing Robot group (Phase II)
- PT (Physical Therapy Only) (Phase II) (Active Comparator): Subjects receive 18 one-hour PT training sessions over 9 weeks. Subjects perform over-ground mobility tasks of increasing challenge with therapist assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Interventions: Other: Physical Therapy Only (Phase II)
- X-PTR, Cross over group for Physical Therapy n Sub-Acute group. (Experimental): Participants enrolled in the physical therapy only group will be given the option to re-enroll as a cross over participant to receive 18 one-hour PT training sessions over 9 weeks while wearing the robot initially parameterized to individual deficit severity. Subjects perform over-ground mobility tasks of increasing challenge with robotic assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Interventions: Device: Cross over group for Physical Therapy n Sub-Acute group. (Phase II)
- C-PTR, Chronic Stroke Subjects to receive robotic gait training therapy. (Experimental): Chronic stroke subjects receive 18 one-hour PT training sessions over 9 weeks while wearing the robot initially parameterized to individual deficit severity. Subjects perform over-ground mobility tasks of increasing challenge with robotic assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Interventions: Device: Chronic Stroke Subjects to receive robotic gait training therapy.

INTERVENTIONS:
Device: PTR Physical Therapy while wearing Robot group (Phase II) — Subjects receive 18 one-hour PT training sessions over 9 weeks while wearing the robot initially parameterized to individual deficit severity. Subjects perform over-ground mobility tasks of increasing challenge with robotic assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Other Names: PTR
  Arms: PTR (Physical Therapy while wearing Robot group) (Phase II)
Other: Physical Therapy Only (Phase II) — Subjects receive 18 one-hour PT training sessions over 9 weeks. Subjects perform over-ground mobility tasks of increasing challenge with therapist assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Other Names: PT
  Arms: PT (Physical Therapy Only) (Phase II)
Device: Cross over group for Physical Therapy n Sub-Acute group. (Phase II) — Participants enrolled in the physical therapy only group will be given the option to re-enroll as a cross over participant to receive 18 one-hour PT training sessions over 9 weeks while wearing the robot initially parameterized to individual deficit severity. Subjects perform over-ground mobility tasks of increasing challenge with robotic assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Other Names: X-PTR
  Arms: X-PTR, Cross over group for Physical Therapy n Sub-Acute group.
Device: Chronic Stroke Subjects to receive robotic gait training therapy. — Chronic stroke subjects receive 18 one-hour PT training sessions over 9 weeks while wearing the robot initially parameterized to individual deficit severity. Subjects perform over-ground mobility tasks of increasing challenge with robotic assist, as needed. Training is generally divided into 3 phases based on individual ability to address gait deficits, postural transitions, physical demand and environmental terrain.
  Other Names: C-PTR
  Arms: C-PTR, Chronic Stroke Subjects to receive robotic gait training therapy.

SUMMARY:
The randomized study (in Phase II of the U44) compares the efficacy and durability of 9 weeks (18 sessions) of robot-assisted physical therapy (PTR) versus physical therapy (PT) alone on foot drop as assessed by gait biomechanics (ankle angle at initial contact, peak swing ankle angle, number of heel-first strikes - % total steps, gait velocity) and blinded clinician assessment (dorsiflexion active range of motion, ankle muscle strength, assistive device needs).

DETAILED DESCRIPTION:
This proposal investigates a portable ankle robot (AMBLE) to be used during over-ground mobility training to reduce foot drop and improve walking function in hemiparetic (half-body, partially paralyzed stroke patients with foot drop (inability to properly lift and clear the foot during walking. About 30% of stroke survivors are left with permanent ankle weakness that impairs their mobility and increases fall-risk. Currently, stroke survivors with foot drop live with a cane or other assistive device, and often ankle-foot braces (AFOs) for safety. These assistive devices do not reverse or reduce the underlying neurological foot drop problem. Recognizing the crucial role of ankle function in walking and balance, and recognizing that the distal part of the lower extremity often suffers the greatest damage after a human stroke, the investigators have come up with a portable ankle robot as a tool for therapists to help shape recovery of walking.

The AMBLE, and its underlying control system, uses information about how patients are walking from one step to another to assist and shape foot lifting so as to help re- train walking recovery by a process that neuroscientists call motor learning. It is the combination of the partially paralyzed stroke survivor's movement efforts with timely assistance "only as needed" by the robot that investigators and others show is the key to movement recovery after stroke. Thus, the ankle robot is not a crutch, but a learning and measuring device that incrementally "gets out of the way" of the learner to facilitate human robot learning such that the human takes over more of the volitional learning.

The research team at University of Maryland has demonstrated in 4 prior studies using seated and treadmill based robot assisted training using a bulky laboratory robot programmed with a motor learning formula that can improve ankle motor control in both the early and chronic phases of stroke, and this can improve over-ground unassisted walking. A significant proportion of stroke survivors showed session by session recovery of volitional (not assisted by the robot) ankle lifting during walking across 6 weeks of three 30- 45 minute sessions of robot training while walking on a treadmill, even years after their stroke. In fact, it has been found that two weeks of 3 sessions per week ankle robotics training was the time profile for most motor learning recovery to reduce foot drop. This information has informed the design of the study described below.

Previous research was done using a bulky, heavy (~8 lbs), and expensive laboratory robot that only allowed seated or treadmill based training because it was tethered by wires. This greatly limits how it can be used by physical therapists, and is not appropriately configured for ease of use by physical therapists in practice. NextStep Robotics invented and built the ankle robots motor learning programs with a lot of input from physical therapists and other rehabilitation clinicians into a portable lightweight robot that can be used over-ground anywhere with blue tooth controls that also tell the therapist precisely how well the stroke survivors is learning, step by step. It is this new portable ankle robot that is configured for use in practice that investigators seek to test in studies with physical therapists using it fully integrated into their usual outpatient stroke mobility recovery training at University of Maryland Orthopedics and Rehabilitation Institute.

This U44 Award from the National Institute of Neurological Disorders and Stroke (NINDS) is not a typical single phase randomized clinical study, but consists of Phase I that completes commercial design of the robot the first year, followed by Phase II randomized clinical trial across years 2-4 of a finalized commercial version of the ankle robot.

Phase II (following completion of commercial design in Phase I) is a randomized (group assignment by chance), blinded (outcome testing done by technicians unaware of patient group assignment), two arm (2 groups) study that investigates the hypothesis that in subacute (6 weeks to 6 months) stroke subjects with foot drop, AMBLE integrated physical therapy (PTR) consisting of 18 training sessions over nine weeks is more effective than usual physical therapy (PT) to improve foot drop outcomes measured by movement analyses of walking, and by standardized clinical assessments of walking including specific foot drop outcomes as assessed by a certified PT clinician (blinded to treatment assignment), cross checked by blinded review of 2 other clinicians of films of the standardized mobility assessments to provide a consensus impartial judgement. Notably, this Phase II study focuses on sub-acute stroke recovery (6 weeks to 6 months) because it represents a therapeutic window into which conventional outpatient physical therapy is typically front-loaded to optimize outcomes. This phase of stroke rehabilitation is selected to test the AMBLE in real world settings when outpatient physical therapy typically occurs, using a treatment frequency and duration (18 physical therapy sessions across 9 weeks) that is representative of practice in Maryland and most of the United States. If wearing the AMBLE robot during physical therapy in this time-frame reduces foot drop and improves longer term outcomes measured 3 months after all robotics therapy has ended, then the investigators will apply for FDA approval for the first robotics device to actively treat foot drop after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* In the subacute phase of stroke recovery (>6 weeks to <6 months post-stroke) with residual hemiparesis of the lower extremity that includes symptoms of foot-drop. - or - In the chronic phase of stroke recovery (>6 months post-stroke) with residual hemiparesis of the lower extremity that includes symptoms of foot-drop.
* Clear indications of hemiparetic gait by clinical observation

Exclusion Criteria:

* Cardiac history of (a) unstable angina, (b) recent (less than 3 months) myocardial infarction, congestive heart failure (NYHA category II); (c) hemodynamically significant valvular dysfunction
* Hypertension that is a contraindication for routine physical therapy (greater than 160/100 on two assessments).
* Medical History: (a) recent hospitalization (less than 3 months) for severe medical disease, (b) symptomatic peripheral arterial occlusive disease, (c) orthopedic or chronic pain conditions that significantly alter gait function, (d) pulmonary or renal failure (e) active cancer
* History of non-stroke neuromuscular disorder restricting gait.
* Aphasia or cognitive functioning that confounds participation, defined as unable to follow 2 step commands or judgment of the medical officer or therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Angle at Initial Contact | Change from Baseline at both 9 Weeks and at 21 Weeks
  Angle at initial contact averaged across each gait cycle for each subject at a given testing time point.
Swing Dorsiflexion | Change from Baseline at both 9 Weeks and at 21 Weeks
  Peak swing dorsiflexion averaged across each gait cycle for each subject at a given testing time point.
Number of Heel-First Foot Strikes | Change from Baseline at both 9 Weeks and at 21 Weeks
  Number of heel-first foot strikes for each subject at a given testing time point.
Gait Velocity | Change from Baseline at both 9 Weeks and at 21 Weeks
  Average gait velocity (meters/second) for each subject at a given testing time point.

SECONDARY OUTCOMES:
Active range of motion for Dorsiflexion | Change from Baseline at both 9 Weeks and at 21 Weeks
  Active range of motion measured for dorsiflexion by blinded clinician.
Ankle Muscle Strength | Change from Baseline at both 9 Weeks and at 21 Weeks
  Measurement of ankle strength by blinded clinician using the MMT (manual muscle testing)
Number of Participants Using Assistive Devices and Ankle Foot Orthoses | Change from Baseline at both 9 Weeks and at 21 Weeks
  Number of Participants Using Assistive Devices and Ankle Foot Orthoses
Dynamic Gait Index | Change from Baseline at both 9 Weeks and at 21 Weeks
  Assesses gait, balance, and fall risk; ranges from 0-24; higher score is better
Berg Balance Scale | Change from Baseline at both 9 Weeks and at 21 Weeks
  A 14-item objective measure designed to assess static balance and fall risk; ranges from 0-56; higher score is better
Stroke Impact Scale | Change from Baseline at both 9 Weeks and at 21 Weeks
  A self-report questionnaire that evaluates disability and health-related quality of life after stroke.
Activities-Specific Balance Confidence Scale | Change from Baseline at both 9 Weeks and at 21 Weeks
  A self-report measure of balance confidence in performing various activities without losing balance; ranges from 0-1600; higher score is better
CES-D (Center for Epidemiological Studies-Depression) | Change from Baseline at both 9 Weeks and at 21 Weeks
  The Center of Epidemiological Studies-Depression, a 20-item measure that asks to rate how often over the past week the patient experienced symptoms associated with depression; ranges from 0-60; high scores indicating greater depressive symptoms.
NIH Stroke Scale | Change from Baseline at both 9 Weeks and at 21 Weeks
  Tool used to quantify the impairment caused by a stroke, composed of 11 items; ranges from 0-42; higher score indicates greater impairment.
Falls Efficacy Scale | Change from Baseline at both 9 Weeks and at 21 Weeks
  A 16-item self-administered questionnaire designed to assess fear of falling; ranges 16-64; higher score indicates greater fear of falling.
Fatigue Assessment Scale | Change from Baseline at both 9 Weeks and at 21 Weeks
  10-item scale evaluating symptoms of fatigue; ranges from 10-50; higher score indicates greater levels of fatigue.
Modified Ashworth Scale | Change from Baseline at both 9 Weeks and at 21 Weeks
  Measures spasticity in patients; ranges from 0-4; higher score indicates more spasticity/rigidity.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Hennessie, MHA, MBA, Study Director — NextStep Robotics Inc.
Locations (1):
- University of Maryland Rehabilitation & Orthopaedic Institute, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Roy A, Hennessie B, Hafer-Macko C, Forrester LW, Westlake K, Macko RF. Adaptive control ankle robotics training durably improves gait biomechanics in chronic hemiparetic stroke and footdrop. J Neuroeng Rehabil. 2025 Dec 29. doi: 10.1186/s12984-025-01834-2. Online ahead of print. No abstract available. PMID 41462280
- [Derived] Roy A, Hennessie B, Hafer-Macko C, Westlake K, Macko R. Dorsiflexion Specific Ankle Robotics to Enhance Motor Learning After Stroke: A Preliminary Report. Res Sq [Preprint]. 2024 Jun 25:rs.3.rs-4390770. doi: 10.21203/rs.3.rs-4390770/v1. PMID 38978605